CLINICAL TRIAL: NCT03792022
Title: Fully Vaccinated Yet Under-vaccinated: Timeliness and Completeness of Routine Childhood Vaccinations by 2 Years of Age in Nigeria
Brief Title: Timeliness and Completeness of Routine Childhood Vaccinations by 2 Years of Age in Nigeria.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Lifespan Healthcare Resource Limited (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Dr.Ihedioha Emmanuel Chukwunwike, Principal Investigator, Lifespan Healthcare Resource Limited
Other Study IDs: 002
Record Dates: First submitted 2018-12-29; First posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Vaccination Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Adherence to timely vaccine uptake
  Interventions: Behavioral: Adherence to timely vaccine uptake

INTERVENTIONS:
Behavioral: Adherence to timely vaccine uptake — Adherence to timely vaccine uptake

SUMMARY:
The timeliness of routine childhood immunization should be an important component in measuring vaccination coverage rates especially in LMIC countries like Nigeria, yet this is overlooked. This study will determine the age- specific immunization timely uptake rates for the various vaccines covered in the routine childhood immunization and seek out factors that affect timely vaccine uptake among Nigerian children.

DETAILED DESCRIPTION:
This study will determine the extent of timely and complete routine childhood vaccination uptake in Nigeria. The investigators will also seek to understand the factors that influence timely/complete uptake and make recommendations. this study will also determine if the present immunization records system in Nigeria is capable of measuring timely immunization uptake.

ELIGIBILITY:
Inclusion Criteria:

* Received all vaccines Available immunization records

Exclusion Criteria:

* Did not receive all vaccines Non- available immunization records

Ages: 1 Month to 24 Months | Sex: All
Age Groups: Child
Study Population: Vaccination records of children who have attended immunization clinics for the last 24 months.
Sampling Method: Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2019-01-10 (Estimated); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-04-02 (Estimated)

PRIMARY OUTCOMES:
Age specific timely vaccination rate for all vaccines in routine vaccination schedule | 24 months
  The primary outcome measure, age- appropriate immunization is defined as receipt of a scheduled vaccine dose within 30 days of the recommended age. Timeliness will be calculated using child health card data as at 31st December 2018. Descriptive statistics will be produced to describe the characteristics of the sample using frequencies and proportions. Descriptive outcome measures for each dose will be coded as either 'no delay'- age appropriately immunized, delay of 1-6 months' , 'delay greater than 6 months', vaccine received 'acceptably early' (within 30 days prior to when it was due), vaccines received 'too early' (within 30 days prior to when it was due) or vaccine dose not recorded.

IPD SHARING:
Plan to Share IPD: No